CLINICAL TRIAL: NCT02162693
Title: A PhaseⅡb, Randomized, Double-blinded, Clinical Trial of Autologous Adipose Tissue-Derived Mesenchymal Progenitor Cells Therapy for Knee Osteoarthritis
Brief Title: Clinical Trial of Autologous Adipose Tissue-Derived Mesenchymal Progenitor Cells (MPCs) Therapy for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: RenJi Hospital (Other); General Hospital of Chinese Armed Police Force (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBMG-KOA-Ⅱb
Record Dates: First submitted 2014-03-19; First posted 2014-06-13 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal progenitor cells (Experimental): Administrated for intra-articular use of Mesenchymal progenitor cells
  Interventions: Biological: Mesenchymal progenitor cells
- Sodium Hyaluronate (Active Comparator): Administrated for intra-articular use of Sodium Hyaluronate.
  Interventions: Biological: Sodium Hyaluronate

INTERVENTIONS:
Biological: Mesenchymal progenitor cells — Administrated for intra-articular injection
  Arms: Mesenchymal progenitor cells
Biological: Sodium Hyaluronate
  Arms: Sodium Hyaluronate

SUMMARY:
Current medication treatments for KOA aim to relieve inflammation and pain, but they do little to delay or reverse the disease progression and most medications have obvious side effects. When the conservative treatments are useless to patients and joint deformities and joint disfunction, the patients may require surgery. Although surgery of the joints can relieve the pain temporarily, long-term effect (over 10 years) is hard to achieve.

DETAILED DESCRIPTION:
Human adipose-derived mesenchymal progenitor cells (haMPCs) are obtained through a series of procedures: firstly, the fresh adipose tissue is digested with collagenase, filtered, centrifuged and then discard mature adipose cells to obtain adipose tissue-derived nuclear cells also called stromal vascular fraction cells (SVFs). In the end, haMPCs are prepared after being purified andamplified to P2-P5. When induced by specific factors, haMPCs have a potential for multilineage differentiation towards bone, cartilage and fat tissue both in vivo and in vitro. The haMPCs can secrete a number of soluble mediators to stimulate the proliferation of endogenous progenitor cells, to act as nutrients, to be immunosuppressive, to be anti-inflammatory, to prevent fibrosis and promote angiogenesis. The cytokines secreted by haMPCs play a synergic role in restoring the dynamic balance of synthesis and decompositon of cartilage tissue, and finally to repair the impaired cartilage.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is between 18-70 years of age, regardless of gender
2. The subject has a Kellgren-Lawrence grading, as determined by American College of Rheumatology (ACR) criteria for osteoarthritis of the knee, below grade 4
3. The subject or the subject's legally acceptable representative must be willing to participate in the trial, to receive cell therapy and to provide signed and dated informed consent forms

Exclusion Criteria:

1. The subject has an allergic history or is of an allergic constitution
2. The subject has uncontrolled or hard-to-control diseases of heart, liver, kidney or lung
3. The subject has uncontrolled or hard-to-control diseases of cardiovascular or endocrine system
4. The subject has severe infectious diseases or a malignant tumour
5. The subject has coagulation disorders
6. The subject has a BMI of over 30
7. The subject has used traditional Chinese medicine containing anti-inflammatory agents in the 2 weeks preceding the trial
8. The subject has received other intra-articular injections in the 2 months preceding the trial
9. The subject has complications or diseases of: systemic or rheumatoid arthritis, Chondrocalcinosis articular， Hemochromatosis，inflammatory arthropathy，avascular necrosis of femoral head，Paget's disease，hemophilic arthropathy，infectional arthritis，Charcot's disease，villonodular synovitis or synovial chondromatosis
10. The subject tests positive for: HIV, hepatitis virus, syphilis or other infectious diseases
11. The subject has a history of alcoholism, drug abuse, or mental illness
12. The subject has participated in any other clinical trial in the 3 months prior to this trial
13. The subject is pregnant, lactating or is planning to conceive within the next 6 months
14. The subject has any other unsuitable or adverse condition to be determined by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
WOMAC Score(The Western Ontario and McMaster Universities Osteoarthritis Index) | 12 months

SECONDARY OUTCOMES:
Recording of Adverse Events and Serious Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, MD, Principal Investigator — RenJi Hospital; Zhongwen Zhang, MD, Principal Investigator — General Hospital of Chinese Armed Police Force
Locations (2):
- China (2):
  - General Hospital of Chinese Armed Police Force, Beijing
  - Shanghai Renji Hospital, Shanghai

REFERENCES:
- [Derived] Lu L, Dai C, Zhang Z, Du H, Li S, Ye P, Fu Q, Zhang L, Wu X, Dong Y, Song Y, Zhao D, Pang Y, Bao C. Treatment of knee osteoarthritis with intra-articular injection of autologous adipose-derived mesenchymal progenitor cells: a prospective, randomized, double-blind, active-controlled, phase IIb clinical trial. Stem Cell Res Ther. 2019 May 21;10(1):143. doi: 10.1186/s13287-019-1248-3. PMID 31113476